CLINICAL TRIAL: NCT04238000
Title: Cerebellar rTMS Theta Burst for Dual-task Walking in Parkinson's Disease:a Double Blind Cross-over Sham-controlled Study Using Wearing Sensors Technology
Brief Title: Cerebellar rTMS Theta Burst for Dual-task Walking in Parkinson's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione Europea di Ricerca Biomedica Ferb Onlus (Other)
Collaborators: University of Kiel (Other); Università degli Studi di Brescia (Other)
Responsible Party: Principal Investigator, Andrea Pilotto, Parkinson's disease Rehabilitation Centre, Fondazione Europea di Ricerca Biomedica Ferb Onlus
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 19/03
Record Dates: First submitted 2020-01-18; First posted 2020-01-23 (Actual); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: Parkinson; Parkinson Disease; Gait Disorders, Neurologic; Parkinsonism; Gait, Festinating
Keywords: repetitive Transcranial Magnetic stimulation; rTMS; wearing sensors; wearables; step variability; gait variability; gait speed; dual-task; dual-task walking; turning
MeSH Terms: conditions — Parkinson Disease; Gait Disorders, Neurologic; Parkinsonian Disorders | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: Each patient received both rTMS and sham cerebellar stimulation in randomized order in two different sessions, separated by at least 2 weeks. In each session, motor tasks, clinical scales and wearing sensor assessments were tested twice in all patients: at baseline (pre-stimulation) and after rTMS (post-stimulation)
Who Masked: Participant, Investigator
Masking Description: The patient and the examiner who administered the clinical scales were blind to the type of rTMS delivered, which was applied by another blinded experimenter.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Real Stimulation (Active Comparator): Cerebellar Repetitive theta burst stimulation will be performed using a 3 pulses at 50-Hz repeated at a rate of 5-Hz; 20 trains of 10 bursts given with 8-s intervals for a total of 600 pulses. Intensity of rTMS was set at the 80% of Amplitude of Motor Threshold (RMT) obtained in the left motor cortex for each subject.
  Interventions: Device: repetitive transcranial magnetic stimulation
- Sham Stimulation (Placebo Comparator): The rTMS coil stimulation will be applied in the same position of the real stimulation. The Stimulation will be performed like in the real arm with the difference that the coil will be masked and thus will be inactive. The patient will hear the same sound of real stimulation, which will be only functionally inactive but will be completely performed (for the whole time of duration of stimulation)
  Interventions: Device: repetitive transcranial magnetic stimulation

INTERVENTIONS:
Device: repetitive transcranial magnetic stimulation — Cerebellar repetitive theta Burst stimulation will be performed as detailed in the Real arm description

SUMMARY:
Objective of the study:

To test the efficacy of theta burst cerebellar stimulation on dual task walking in Parkinson's disease using a cross-over design and wearing sensors technology

Design:

Twenty Parkinson's disease patients with no dementia will be recruited for a cross-over sham-controlled study. Each patient will undergo a sham stimulation or a single session of cerebellar theta burst stimulation with a wash out period of at least 14 days.

Each patient will be evaluated before and after stimulation by a battery of gait and movement tests using wearing sensors technology .

DETAILED DESCRIPTION:
There are no medical effective treatments for dual-task gait in Parkinson's disease. Imaging, neurophysiology and pathology studies suggested cerebellum as possible target of brain stimulation for dual-task walking for theta Burst repetitive Transcranial magnetic stimulation

Objective of the study:

To test the efficacy of theta burst cerebellar stimulation on gait in Parkinson's disease using a cross-over design and wearing sensors technology

Design:

Parkinson's disease patients able to walk and without dementia/behavioral disturbances will be recruited for a cross-over sham-controlled study. Each patient will undergo a sham stimulation or a single session of cerebellar theta burst stimulation with a wash out period of at least 14 days.

Repetitive cerebellar theta burst stimulation will be performed by Duo-Mag XT100, using a 3 pulses at 50-Hz repeated at a rate of 5-Hz; 20 trains of 10 bursts given with 8-s intervals for a total of 600 pulses. Intensity of rTMS was set at the 80% of Amplitude of Motor Threshold (RMT) obtained in the left motor cortex for each subject.

A sample size of 20 subjects with complete stimulation (2 stimulations per subject, for a total number of stimulation)

Each patient will be evaluated before and after stimulation by a battery of gait and movement tests using wearing sensors technology.

Sensors assessment:

The following gait parameters will be evaluated in normal and cognitive/motor dual-tasks:

i) step length ii) step variability iii) step phases iv) turning speed

ELIGIBILITY:
Inclusion Criteria:

* established Parkinson's disease
* ability to stand alone and walk without support

Exclusion Criteria:

* dementia or behavioral alterations
* contraindication to stimulation

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-04-01 (Estimated); Study Completion 2020-06-01 (Estimated)

PRIMARY OUTCOMES:
Step variability in dual-task walking | Changes from Baseline to immediately after stimulation
  Step variability will be assessed in normal, cognitive/motor dual-task conditions walking
Step length in dual-task walking | Changes from Baseline to immediately after stimulation
  Step length will be assessed in normal, cognitive/motor dual-task conditions
Gait speed in dual-task walking | Changes from Baseline to immediately after stimulation
  Gait speed will be assessed in normal, cognitive/motor dual-task conditions

SECONDARY OUTCOMES:
Turning speed in timed up and go tests | Changes from Baseline to immediately after stimulation
  Turning will be assessed y wearing sensors during timed up and go tests
total distance of dual-task walking | Changes from Baseline to immediately after stimulation
  The total distance of one minute normal/motor/cognitive dual-task walking will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Pilotto, MD, Principal Investigator — FERB Onlus
Locations (1):
- Parkinson's disease Rehabilitation Centre - FERB ONLUS, Trescore Balneario, Italy

IPD SHARING:
Plan to Share IPD: Yes
The whole study will be published in medical journal
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: In the publication, within the next year
Access Criteria: on line availability